CLINICAL TRIAL: NCT02785250
Title: A Phase 1b/2 Study of an Immunotherapeutic Vaccine, DPX-Survivac With Low Dose Cyclophosphamide and Epacadostat (INCB024360) in Patients With Recurrent Ovarian Cancer
Brief Title: Study of DPX-Survivac Therapy in Patients With Recurrent Ovarian Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ImmunoVaccine Technologies, Inc. (IMV Inc.) (Industry)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONC-DPX-Survivac-06; DeCidE1 (Other: Sponsor)
Record Dates: First submitted 2016-05-18; First posted 2016-05-27 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Recurrent Epithelial Ovarian Cancer; Recurrent Fallopian Tube Cancer; Recurrent Peritoneal Cancer
Keywords: T cell activation; immunotherapy; ovarian; fallopian tube; peritoneal; cancer; recurrent; tumor; measurable
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Neoplasms; Recurrence | interventions — Cyclophosphamide; epacadostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): DPX-Survivac, Cyclophosphamide, Epacadostat (Phase 1 and initially Phase 2)
  Interventions: Other: DPX-Survivac; Drug: Cyclophosphamide; Drug: Epacadostat (INCB024360)
- Arm 2 (Experimental): DPX-Survivac, Cyclophosphamide (in Phase 2 only)
  Interventions: Other: DPX-Survivac; Drug: Cyclophosphamide

INTERVENTIONS:
Other: DPX-Survivac — SubQ injection
Drug: Cyclophosphamide — PO BID
Drug: Epacadostat (INCB024360) — PO BID
  Arms: Arm 1

SUMMARY:
T cell activating therapy DPX-Survivac, low dose oral cyclophosphamide, and IDO1 inhibitor epacadostat will be tested together for the first time in patients with recurrent ovarian, fallopian tube, or peritoneal cancer to determine the safety and potential immune-modulating activity of the combination of these agents.

DETAILED DESCRIPTION:
The Phase 1b component is a multicenter, non-randomized, open label, uncontrolled, safety and effectiveness study to identify the recommended Phase 2 dose (R2PD) of epacadostat in combination with DPX-Survivac and cyclophosphamide.

The Phase 2 component was initially a multicenter, randomized, open-label study to evaluate the safety and effectiveness of DPX-Survivac + cyclophosphamide with or without the RP2D of epacadostat. The design of the study has been amended to a single arm study in which up to 16 evaluable subjects will be enrolled to received DPX-Survivac plus intermittent low dose cyclophosphamide (i.e. treatment arm 2).

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed, stage IIc-IV epithelial ovarian, fallopian tube or peritoneal cancer
* Platinum-resistant or -sensitive subjects after completing first-line treatment (debulking surgery and adjuvant or neoadjuvant treatment with standard of care treatment such as carboplatin and paclitaxel). Subjects may have had any number of subsequent lines of chemotherapy.
* Must have evidence of progressive disease with either biochemical (i.e. rising CA-125) and/or radiologic progression
* Must have measurable disease by RECIST v1.1, a successful pre-treatment tumor biopsy, and be willing to undergo tumor biopsy during treatment
* Ambulatory with an ECOG 0-1
* Life expectancy ≥ 6 months
* Meet protocol-specified laboratory requirements

Key Exclusion Criteria:

* Eligible for otherwise curative treatment or undergoing concurrent therapy
* Prior receipt of survivin based vaccines or immune checkpoint inhibitors (e.g. anti-CTLA-4, anti-PD-1, anti-PD-L1, or any other antibody or drug specifically targeting T cell co-stimulation) or an IDO inhibitor
* Concurrent second malignancy other than non-melanoma skin cancer, cervical carcinoma in situ, or controlled bladder cancer
* Clinical ascites
* Any single lesion greater than or equal to 4 cm (per RECIST v1.1)
* Malignant bowel obstruction
* History of autoimmune disease requiring treatment within the last two years (except vitiligo or diabetes)
* Recent history of thyroiditis
* Presence of a serious acute infection or chronic infection
* Active central nervous system (CNS) or leptomeningeal metastasis (brain metastases)
* GI condition that might limit absorption of oral agents
* Other serious intercurrent chronic or acute illness, including myocardial infarction or cerebrovascular event within 6 months
* Ongoing treatment with steroid therapy or other immunosuppressive
* Receipt of monoamine oxidase inhibitors (MAOIs) or UGT1A9 inhibitors
* Receipt of live attenuated vaccines
* Acute or chronic skin and/or microvascular disorders
* Edema or lymphedema in the lower limbs > grade 2

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2016-04; Primary Completion 2020-10 (Actual); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Safety as measured by adverse event reporting (CTCAE) | up to 13 months
Objective Response Rate (Phase 2 only) | up to 13 months
  Evaluated using modified RECIST v1.1

SECONDARY OUTCOMES:
Objective Response Rate (for each treatment group) | up to 13 months
  Evaluated using modified RECIST v1.1
Duration of Response | up to 13 months
Cell mediated immunity as measured by the antigen specific response in peripheral blood | bimonthly for up to 13 months
Evaluation of treatment-induced changes in tumor infiltrating lymphocytes | at 8 to 10 weeks
Time to Progression | up to 13 months
Overall Survival | up to 13 months

CONTACTS AND LOCATIONS:
Locations (9):
- United States (6):
  - Stanford University, Palo Alto, California
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Lenox Hill Hospital, New York, New York
  - Oregon Health & Sciences University, Knight Cancer Institute, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Mary Crowley Cancer Research Center, Dallas, Texas
- Canada (3):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Princess Margaret Hospital, Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec